CLINICAL TRIAL: NCT02900885
Title: Study of Ocular Torsion in Patients Suffering From Palsy of the Superior Rectus Extraocular Muscle
Acronym: EXCYCLO
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: NI_VTN_2015_1
Record Dates: First submitted 2016-09-06; First posted 2016-09-14 (Estimated); Last update posted 2016-09-14 (Estimated); Status verified 2016-09

CONDITIONS: Superior Rectus Palsy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

SUMMARY:
Retrospective medical chart and medical imaging file review of patients suffering from palsy of the superior rectus extraocular muscle

ELIGIBILITY:
Inclusion Criteria:

* Patient with unilateral muscular palsy of the superior rectus muscle
* Patient must have a binocular vision as characterized by Lang test

Exclusion Criteria:

* bilateral impairment of the superior rectus muscle
* presence of an orbital lesion (orbital trauma, tumor or pseudo-tumor)
* thyroid orbitopathy
* No binovular vision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patiente suffering from unilateral muscular palsy of the superior rectus extraocular muscle
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2012-01; Primary Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Excyclotorsion of the eye as measured in angle degrees by retinophotography | Within 1 week prior to corrective surgery